CLINICAL TRIAL: NCT04173247
Title: Pilot Study of KeraStat® Cream for Radiation Dermatitis During Head and Neck Radiotherapy
Brief Title: Study of KeraStat Cream for Radiation Dermatitis During Head and Neck Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: KeraNetics, LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00062012; WFBCCC 97319 (Other: IRB - Wake Forest University Health Science); P30CA012197 (NIH)
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Results first posted 2023-09-07 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Cancer; Radiation Dermatitis
MeSH Terms: conditions — Head and Neck Neoplasms; Radiodermatitis | interventions — eucerin; Gels; cetyl alcohol, propylene glycol, sodium lauryl sulfate non-lipid cleansing lotion; Zinc Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- KeraStat Skin Cream Arm (Experimental): Patients randomized to the KeraStat arm will be provided with KeraStat Skin Cream for application as often as needed but at least twice daily, morning and evening using the product on the start date of radiation and continue until returning for follow up approximately one month after last radiation treatment.
  Interventions: Device: KeraStat Cream
- Routine Skin Care Arm (RSC Arm) (Active Comparator): Patients randomized to this arm will apply commercially available products from a list provided at least twice daily using the product on the start date of radiation and continue until returning for follow up approximately one month after last radiation treatment.
  Interventions: Other: Routine Skin Care - Commercially Available Agents

INTERVENTIONS:
Device: KeraStat Cream — KeraStat Cream is a non-sterile, non-implantable, emollient-based wound dressing intended to act as a protective covering in the management of a variety of skin conditions.
  Arms: KeraStat Skin Cream Arm
Other: Routine Skin Care - Commercially Available Agents — Commercially available skin moisturizers from an approved list that do not interfere with radiation.
  Other Names: Aveeno Skin Relief lotion; Eucerin; Lubriderm; Calendula cream or gel; Aloe vera gels; Cetaphil; CeraVe; Petroleum based with mineral oil ointments: Aquaphor, Balmex, Elta
  Arms: Routine Skin Care Arm (RSC Arm)

SUMMARY:
This is a single site, randomized, open-label comparison pilot study to assess the feasibility and effectiveness of KeraStat Cream compared with routine skin care (RSC) in managing radiotherapy-induced early adverse skin reaction (EASR) in patients undergoing radiotherapy to the head and/or neck.

Hypothesis: The use of KeraStat Cream in patients receiving radiotherapy for head and neck is feasible, tolerable, and reduces the severity of early adverse skin reaction in the treated region of interest.

DETAILED DESCRIPTION:
Primary Objective(s)

• To determine the feasibility of the use of KeraStat Cream in patients receiving radiotherapy for head and neck cancer.

Secondary Objective(s)

* To determine the tolerability of KeraStat Cream in patients receiving radiotherapy for head and neck cancer compared to routine skin care.
* To assess the effectiveness of KeraStat Cream in reducing the severity of EASR in patients receiving radiotherapy for head and neck cancer, compared to routine skin care. This will be performed by evaluating:
* Objective evaluation of EASR using the CTCAE Version 5.0 scale of radiation dermatitis,
* Patient-reported outcomes of radiation dermatitis using the PRO-CTCAE version 1.0, and
* Dermatologic-specific quality of life assessment
* To estimate the amount of KeraStat Cream used per patient and coverage on the skin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of head and neck cancer planned to receive conventionally-fractionated definitive radiotherapy to the head and neck to a total prescribed dose of at least 60 Gy
* Able and willing to sign protocol consent form
* Able and willing to complete tolerability and quality of life assessments
* Able and willing to have photographs of the affected area taken regularly

Exclusion Criteria:

* Women who are pregnant, lactating/nursing or plan to become pregnant
* Previous radiation therapy to the area to be treated with radiation therapy
* Active, medically necessary use of topical corticosteroids in the irradiation area
* Active scleroderma or lupus requiring systemic medication
* Treatment with anti-EGFR antibodies for head and neck cancer (previously or planned)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Hughes, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | KeraStat Skin Cream Arm | Routine Skin Care Arm (RSC Arm)
Started | 14 | 14
Completed | 12 | 12
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Death | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KeraStat Skin Cream Arm | Routine Skin Care Arm (RSC Arm) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Median (Full Range); unit: years] | 63.5 [30 to 77] | 64.5 [47 to 78] | 64 [30 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 11 | 7 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 11 | 21
  Black | 1 | 1 | 2
  Other | 0 | 0 | 0
  Unknown | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Completion Rate of Use of KeraStat Cream
Description: Feasibility of use of KeraStat Cream is measured by participant compliance with an average of 10 or more applications per week being classified as complaint. In each arm, a 95% confidence interval will be calculated around the estimate of compliance.
Time Frame: Up to 1 month post treatment with radiation therapy (6-7 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | KeraStat Skin Cream Arm | Routine Skin Care Arm (RSC Arm)
Number analyzed (Participants) | 12 | 12
Participants | 10 | 7

2. Secondary Outcome: Number of Participants Discontinuing Skin Care Regimen
Description: Tolerability is measured by the number of patients who discontinue skin care regimen due to intolerance for any reason. In each arm, a 95% confidence interval will be calculated around the estimate of tolerability.
Time Frame: Up to 1 month post treatment with radiation therapy (6-7 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | KeraStat Skin Cream Arm | Routine Skin Care Arm (RSC Arm)
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

3. Secondary Outcome: Number of Participants With Grade 2+ Radiation Dermatitis
Description: Objective assessment of early adverse skin reaction defined as Grade 2+ using the CTCAE version 5.0 scale of radiation dermatitis will be compared between the KeraStat group and the RSC group at the end of treatment, using a Fisher's exact test.
Time Frame: Up to 1 month post treatment with radiation therapy (6-7 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | KeraStat Skin Cream Arm | Routine Skin Care Arm (RSC Arm)
Number analyzed (Participants) | 12 | 12
Participants | 9 | 7

4. Secondary Outcome: Number of Participants Reporting Radiation Skin Reaction
Description: Patient-reported assessment of skin toxicity using the PRO-CTCAE version 1.0 scale of radiation skin symptoms (skin dryness, itching, radiation skin reaction and skin darkening). Score scale is none to very severe and Yes or No for skin darkening.
Time Frame: Up to 1 month post treatment with radiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | KeraStat Skin Cream Arm | Routine Skin Care Arm (RSC Arm)
Number analyzed (Participants) | 12 | 12
Participants | 8 | 10

5. Secondary Outcome: Dermatology Life Quality Index Questionnaire
Description: A 10-item questionnaire to measure how skin problems have affected participants' lives. Scoring for each question ranges from 0-3 with very much scored as 3 and not at all or not relevant score as 0. The DLQI is calculated by summing the score of each questions resulting in a maximum score of 30 and a minimum score of 0. The higher the score, the more quality of life is impaired. The mean of the highest DLQI score across all time points will be compared between the KeraStat and RSC groups using a t-test.
Time Frame: At weeks 1-6 and up to 1 month post treatment with radiation therapy
Population: Dlqi scores below are averaged over weeks 1-6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | KeraStat Skin Cream Arm | Routine Skin Care Arm (RSC Arm)
Number analyzed (Participants) | 12 | 12
units on a scale | 1.5 (2.5) | 1.9 (2.5)
Statistical Analysis 1: Comparison: KeraStat Skin Cream Arm vs Routine Skin Care Arm (RSC Arm); Test type: Other — A t-test with 180 degrees of freedom to compare the mean DLQI score over the 6 weeks in arm1 to the mean DLQI score over six weeks in arm2; p = 0.28, t-test, 1 sided

6. Secondary Outcome: Number of Tubes of KeraStat Cream Used to Calculate Skin Coverage
Description: Skin coverage is defined as the total number of tubes of KeraStat Cream used over 7 weeks OVER ALL participants in the KeraStat arm only.
Time Frame: Up to 1 month post treatment with radiation therapy (7 weeks)
Population: Number of tubes over 7 weeks, in KeraStat arm only
Measure: Number; unit: total number of tubes of KeraStat used
Arm/Group | KeraStat Skin Cream Arm | Routine Skin Care Arm (RSC Arm)
Number analyzed (Participants) | 12 | 0
total number of tubes of KeraStat used | 49 |

ADVERSE EVENTS:
Time Frame: Up to 1 month post treatment with radiation therapy (6-7 weeks)
Arm/Group | KeraStat Skin Cream Arm | Routine Skin Care Arm (RSC Arm)
All-Cause Mortality (participants affected / at risk) | 1/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 3/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KeraStat Skin Cream Arm (N=12) | Routine Skin Care Arm (RSC Arm) (N=12)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KeraStat Skin Cream Arm (N=12) | Routine Skin Care Arm (RSC Arm) (N=12)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT04173247/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT04173247/ICF_000.pdf